CLINICAL TRIAL: NCT03019159
Title: Efficacy and Cost-effectiveness Assessment of a Follow-up With Tele-consulting for Patients With Chronic Renal Failure Under Peritoneal Dialysis
Brief Title: Assessment of a Follow-up With Tele-consulting for Patients With Renal Failure Under Peritoneal Dialysis
Acronym: HSMDP
Status: Withdrawn | Type: Observational
Why Stopped: Support funding of the regional health authority stopped
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Agence Regionale de Sante d'Ile de France (Other Government)
Responsible Party: Sponsor
Other Study IDs: TLM-HSMDP
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Renal Failure; Peritoneal Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tele-consulting: One visit out of two takes place with teleconsulting and the other is a face-to-face consultation
  Interventions: Device: Teleconsulting
- No tele-consulting

INTERVENTIONS:
Device: Teleconsulting
  Other Names: Telemedicine
  Groups: Tele-consulting

SUMMARY:
The objective of the study is to determine whether tele-consulting for the follow up of patients with renal failure under peritoneal dialysis would not increase the risk of experiencing a severe adverse event

ELIGIBILITY:
Inclusion Criteria:

* Patient under peritoneal dialysis for more than three month
* Patient thought to be able to perform peritoneal dialysis alone or with the help of health care professionnals
* Patients or health care professionnals thought to be able to use telemedicine

Exclusion Criteria:

* No DSL Network
* No GSM Network
* Patients who can not express their opposition to the participation to this study because of limited mental abilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with renal failure under peritoneal dialysis
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Severe adverse events | Within 2 years after enrollment
  Death, Peritonitis, acute pulmonary edema, symptomatic hyperkalemia or with EKG signs, severe and resistant hypertension, with uremia > 40 mmol/L

SECONDARY OUTCOMES:
Number of hospitalisations | Within 2 years after enrollment
Number of consultations | Within 2 years after enrollment
Number of sanitary transportation | Within 2 years after enrollment
Mean length of hospital stay | Within 2 years after enrollment
Global costs | 6 months after the first patient enrollment
Patients satisfaction | 1 year after enrollment
Satisfaction of the professionnals | 6 months after enrollment of the first patient

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Roueff, MD, Principal Investigator — Pôle CTIRC. Hôpitaux Saint Maurice; Isabelle Durand-Zaleski, MD, PhD, Principal Investigator — DRCD URC Eco. Assistance Publique - Hôpitaux de Paris
Locations (1):
- CTIRC - Hôpitaux Saint Maurice, Saint-Maurice, France

REFERENCES:
- [Background] Gallar P, Vigil A, Rodriguez I, Ortega O, Gutierrez M, Hurtado J, Oliet A, Ortiz M, Mon C, Herrero JC, Lentisco C. Two-year experience with telemedicine in the follow-up of patients in home peritoneal dialysis. J Telemed Telecare. 2007;13(6):288-92. doi: 10.1258/135763307781644906. PMID 17785025
- [Background] Kidholm K, Ekeland AG, Jensen LK, Rasmussen J, Pedersen CD, Bowes A, Flottorp SA, Bech M. A model for assessment of telemedicine applications: mast. Int J Technol Assess Health Care. 2012 Jan;28(1):44-51. doi: 10.1017/S0266462311000638. PMID 22617736